CLINICAL TRIAL: NCT02837562
Title: Risk of Radiation-induced Cataracts Among Interventional Cardiology Staff- CATaracts Attributed to Radiation in the CaTh Lab: The IC-CATARACT Study
Brief Title: Risk of Radiation-induced Cataracts Among Interventional Cardiology Staff
Acronym: IC-CATARACT
Status: Withdrawn | Type: Observational
Why Stopped: 0
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Dallas VA Research Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: STU-042016-016
Record Dates: First submitted 2016-06-24; First posted 2016-07-19 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Cataract
Keywords: Radiation exposure; Cardiac catheterization
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Interventional Cardiology/Cath Lab Staff: This is considered to be the "case" or group under study. These are Interventional Cardiology/ Cardiac Cath lab staff that are exposed to radiation as a result of their role as Cardiac Cath lab staff.
  Intervention: Slit lamp eye examination
  Interventions: Other: Slit lamp eye examination
- Non-Interventional Cardiology/ Controls: This is considered to be the "control" or comparison group. These are non-interventional cardiology/ non-cardiac cath lab staff that are not exposed to radiation as they do no operate/ work in the Cardiac Cath Lab.
  Intervention: Slit lamp eye examination
  Interventions: Other: Slit lamp eye examination

INTERVENTIONS:
Other: Slit lamp eye examination — All participants in the trial will undergo a slit lamp eye examination

SUMMARY:
The goal of the present study is to evaluate the prevalence of radiation-associated lens opacities among interventional cardiology staff members (such as physicians, technicians, and nurses) and determine its association with occupational history.

The hypothesis of the study is that interventional cardiology staff will have high prevalence of radiation-induced lens opacities, which will be higher than non-interventional cardiology staff and will correlate with the estimated cumulative lifetime dose.

DETAILED DESCRIPTION:
This is an observational, cross-sectional study to evaluate the prevalence of posterior subcapsular cataract (PSC) and its association with prior occupational history of radiation exposure. Participants of the Society of Cardiovascular Angiography and Interventions 2016 Scientific Sessions to be held in Orlando, FL May 4th to May 7th, will be invited to participate. Both interventional cardiology and non-interventional cardiology staff and non-clinical participants will be assessed. Written informed consent will be obtained from all participants. They will subsequently be asked to complete a questionnaire on occupational radiation exposure, workplace practices and medical history followed by dilated slit lamp examination using a modified Merriam-Focht scoring system.

ELIGIBILITY:
Inclusion Criteria:

* Willing to undergo eye examination
* Participant at Society of Cardiovascular Angiography and Interventions 2016 Scientific Sessions

Exclusion Criteria:

* Known pre-existing severe eye disease, such as glaucoma
* Prior lens surgery
* Known hypersensitivity to the mydriatic agents
* Any other conditions that may preclude participation/ performance of slit lamp eye examination/ use of mydriatics, in the opinion of the investigator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants of the Society of Cardiovascular Angiography and Interventions (SCAI) 2016 Scientific Sessions to be held in Orlando, FL May 4th to May 7th, 2016
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Radiation associated lens opacities | At study completion, approximately 30 minutes after administration of mydriatic eye drops
  Measured by slit-lamp eye examination

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No